CLINICAL TRIAL: NCT07344948
Title: A First in Human, Phase 1/1b Study of Single and Multiple Ascending Dosing Administration of NTX110253 in Healthy Participants and Participants With Stable Schizophrenia
Brief Title: Single and Multiple Ascending Doses of NTX-253 in Healthy Participants and Participants With Stable Schizophrenia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Neurosterix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTX-0253-101
Record Dates: First submitted 2025-11-14; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; Schizophrenia Diagnosis
Keywords: Phase 1; Healthy volunteer; Schizophrenia; Pharmacokinetics; Single ascending dose; Multiple ascending dose; Food effect; Safety
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Crossover design for fasted/fed cohort
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- NTX-253 Part 1a (Experimental): Participants will be assigned to receive one of multiple single ascending daily oral doses of NTX-253
  Interventions: Drug: NTX-253
- Placebo Part 1a (Experimental): Participants will be assigned to receive one of multiple single ascending daily oral doses of placebo
  Interventions: Drug: Placebo
- NTX-253 Part 1b (Experimental): Participants will receive the maximum tolerated single oral dose of NTX-253
  Interventions: Drug: NTX-253
- NTX-253 Part 2 (Experimental): Participants will be assigned to receive one of multiple ascending oral daily doses of NTX-253 for 10 days
  Interventions: Drug: NTX-253
- Placebo Part 2 (Experimental): Participants will be assigned to receive one of multiple ascending daily oral doses of placebo for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NTX-253 — Oral Capsule
  Arms: NTX-253 Part 1a; NTX-253 Part 1b; NTX-253 Part 2
Drug: Placebo — Oral capsule
  Arms: Placebo Part 1a; Placebo Part 2

SUMMARY:
This study will assess the safety, tolerability, and pharmacokinetics of NTX-253 following oral administration in both healthy adult participants as well as adult participants with stable schizophrenia.

DETAILED DESCRIPTION:
This study will assess the safety, tolerability, and pharmacokinetics of NTX-253 following oral administration in both healthy adult participants as well as adult participants with stable schizophrenia. NTX-253 is an investigational drug being developed for the treatment of schizophrenia. The study will consist of a single ascending dose (SAD - Part 1a) phase which will include a food effect cohort, and a cerebrospinal fluid (CSF - Part 1b) cohort in healthy volunteers. Participants will receive a single dose of either oral NTX-253 or placebo. The multiple ascending dose (MAD - Part 2) phase will follow. In Part 2, participants will be dosed for 10 consecutive days with either NTX-253 or placebo. Each phase will include sequential escalating doses in healthy volunteers. Two cohorts in the MAD phase will include stable schizophrenic adult participants who have had antipsychotic medication withdrawn for up to 8 days prior to dosing with NTX-253.

ELIGIBILITY:
Primary Inclusion Criteria:

* Male or non-pregnant, non-lactating female participants, ages 18-55 who are not of childbearing potential, with a truly abstinent lifestyle, or agrees to use medically acceptable forms of birth control
* Part 1 a/b, Part 2 Cohort 7 only: Body mass index (BMI) within the range ≥18.0 to ≤30.0 kg/m2
* Participants in the food effect cohort must be willing to eat a single high fat breakfast
* (Part 2 only): Stable schizophrenia participants (schizophrenia cohorts only)
* Body mass index (BMI) within the range ≥17.5 to ≤36.0 kg/m2
* Positive and Negative Syndrome Scale (PANSS) total score <80 at screening

Primary Exclusion Criteria:

* (Part 1a/b, Part 2 Healthy): History of or current clinically significant medical or mental illness
* Cancer diagnosis/treatment in the past 7 years
* Acute or chronic gastrointestinal conditions that would interfere with drug tolerance or absorption
* Any clinically significant, abnormal 12 lead ECG
* Part 2: Any primary DSM-5TR disorder other than schizophrenia
* Participants with schizophrenia who are considered resistant/refractory to antipsychotic treatment by history; history of clozapine use.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of reported Adverse Events | From baseline until Day 8 after a single dose, Day 17 (healthy volunteers) or Day 35 (participants with stable schizophrenia).
  Safety and tolerability will be assessed by the incidence and severity of treatment-emergent adverse events.
Number of Adverse Events of Special Interest (AESI) | From baseline until Day 8 after a single dose, Day 17 (healthy volunteers) or Day 35 (participants with stable schizophrenia).
  Safety and tolerability will be assessed by the incidence and severity of AESIs.
Number of dose limiting treatment emergent adverse events (TEAE) | From baseline until Day 8 after a single dose, Day 17 (healthy volunteers) or Day 35 (participants with stable schizophrenia).
  Safety and tolerability will be assessed by the incidence and severity of serious or dose limiting TEAEs.
Vital Signs: Change in blood pressure | From baseline until Day 8 after a single dose, Day 17 (healthy volunteers) or Day 35 (participants with stable schizophrenia).
  Blood pressure measurements
Vital Signs: Change in temperature | From baseline until Day 8 after a single dose, Day 17 (healthy volunteers) or Day 35 (participants with stable schizophrenia).
  Oral temperature measurement
Vital Signs: Change in respiratory rate | From baseline until Day 8 after a single dose, Day 17 (healthy volunteers) or Day 35 (participants with stable schizophrenia).
  Respiratory rate (number of breaths per minute) measurements
Vital Signs: Change in heart rate | From baseline until Day 8 after a single dose, Day 17 (healthy volunteers) or Day 35 (participants with stable schizophrenia).
  Pulse measurements.
Change in physical examination | From baseline until Day 8 after a single dose, Day 17 (healthy volunteers) or Day 35 (participants with stable schizophrenia).
  Investigator will perform complete physical exam and document any clinically significant conditions.
Clinical Laboratory Tests | From baseline until Day 8 after a single dose, Day 17 (healthy volunteers) or Day 35 (participants with stable schizophrenia).
  Hematology, serum chemistry, urinalysis, and coagulation tests.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) [Pharmacokinetics] | From baseline until up to 168 hours after a single dose, or until up to 168 hours after the last dose in the multiple dose cohorts.
  Samples will be collected periodically until:
  * 72 hours after a single dose with optional samples collected at 96, 120, 144, and 168 post-dose.
  * 72 hours after multiple doses with optional samples collected at 96, 120, 144, and 168 hours after the last dose.
Time of Cmax (tmax) [Pharmacokinetics] | From baseline until up to 168 hours after a single dose, or until up to 168 hours after the last dose in the multiple dose cohorts.
  Samples will be collected periodically until:
  * 72 hours after a single dose with optional samples collected at 96, 120, 144, and 168 post-dose.
  * 72 hours after multiple doses with optional samples collected at 96, 120, 144, and 168 hours after the last dose.
Apparent terminal half-life (t1/2) | From baseline until up to 168 hours after a single dose, or until up to 168 hours after the last dose in the multiple dose cohorts.
  Samples will be collected periodically until:
  * 72 hours after a single dose with optional samples collected at 96, 120, 144, and 168 post-dose.
  * 72 hours after multiple doses with optional samples collected at 96, 120, 144, and 168 hours after the last dose.
Amount of unchanged drug excreted in urine (Ae) [urinary excretion) | From baseline until 72 hours after a single dose, or until the last dosing on Day 10 in the multiple dose cohort.
  Samples will be collected in select cohorts from baseline until 72 hours after a single dose, or at baseline and on the last dosing day after multiple dose administrations.
Percent of dose excreted as unchanged drug in urine (Ae%) [urinary excretion] | From baseline until 72 hours after a single dose, or until the last dosing on Day 10 in the multiple dose cohort.
  Samples will be collected in select cohorts from baseline until 72 hours after a single dose, or at baseline and on the last dosing day after multiple dose administrations.
Renal clearance (Clr) [urinary excretion] | From baseline until 72 hours after a single dose, or until the last dosing on Day 10 in the multiple dose cohort.
  Samples will be collected in select cohorts from baseline until 72 hours after a single dose, or at baseline and on the last dosing day after multiple dose administrations.
Maximum observed CSF concentration (Cmax, CSF) [Pharmacokinetics] | From baseline until 12 hours after a single dose.
  CSF samples will be collected at periodic intervals until 12 hours after a single dose in a single dose CSF cohort.
Time corresponding to Cmax (Tmax, CSF) [Pharmacokinetics] | From baseline until 12 hours after a single dose.
  CSF samples will be collected at periodic intervals until 12 hours after a single dose in a single dose CSF cohort.
QT/QTc potential interval prolongation and plasma concentration | From baseline until 72 hours post-dose in the single dose cohorts, then from baseline until Day 13 in the multiple dose cohorts.
  Electrocardiograms (ECGs) will be collected to assess the potential for QT/QTc interval prolongation and ΔQTc as measured by:
  • Change from baseline in cardiac measurements

CONTACTS AND LOCATIONS:
Overall Officials: Doug Feltner, MD, Study Director — Neurosterix
Locations (1):
- Collaborative Neuroscience Research, LLC - CenExel, Los Alamitos, California, United States

IPD SHARING:
Plan to Share IPD: No